CLINICAL TRIAL: NCT01292122
Title: A Single-Center, Prospective, Randomized Study of VCT-01™ in Split-Thickness Skin Graft Donor Site Wounds
Brief Title: Safety Study of VCT-01™ in Split-Thickness Skin Graft Donor Site Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-GDS-001-VCT
Record Dates: First submitted 2011-01-28; First posted 2011-02-09 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Wounds
Keywords: Wounds; Grafts; Wound Healing; Cell Therapy; Split-thickness skin graft donor site wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VCT-01-treated STSG donor site wound (Experimental): Application of VCT-01 to STSG donor site wound at Day 0
  Interventions: Device: VCT-01

INTERVENTIONS:
Device: VCT-01 — Application of bi-layered living cell-based product (VCT-01) to STSG donor site wound at Day 0

SUMMARY:
The purpose of this study is to evaluate the safety of VCT-01 in split-thickness skin graft (STSG) donor site wounds and assess selected parameters of healing at the VCT-01-treated donor site.

DETAILED DESCRIPTION:
An initial cohort of 5 subjects will be allocated to Group A. When all subjects enrolled in Group A have completed 14 days of post-treatment follow-up, results of donor site evaluations, histological analyses and reported adverse events will be reviewed by the Investigator and study Sponsor. If the data is suggestive of clinical benefit following treatment and absent any serious and/or unexpected adverse events, which are, in the opinion of the investigator, related to the treatment, the remaining subjects will be enrolled and randomized to Groups B, C or D.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age but no more than 55 years of age.
2. Subject has a primary wound which requires treatment with a split-thickness skin graft; the graft cannot be harvested from a site from which a skin graft was previously obtained. If the primary wound is a result of a thermal or chemical burn, the total body surface area must be less than 15%.
3. Females of childbearing potential must have a documented negative urine pregnancy test and must agree to use highly effective contraceptives for 6 months post-treatment.
4. Subject has read, understood and signed a Health Research Ethics Board-approved Informed Consent Form.
5. Subject is able and willing to comply with study procedures and instructions.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. Clinically significant disease or condition that may compromise graft take and/or donor site healing (e.g. the presence of a bleeding disorder, capillary fragility, venous or arterial disorder directly affecting the donor site to be treated, known or suspected systemic malignancies, human immunodeficiency virus infection, renal or liver disease, uncontrolled diabetes mellitus, thrombocytopenia, vasculitis, poor nutritional status).
3. Subjects who are currently receiving or have received within two months prior to treatment: systemic, inhaled or intranasal corticosteroids or immunosuppressant agents. Subjects receiving therapeutic doses of anticoagulants for pre-existing medical conditions (e.g. Plavix, Coumadin, Heparin, low molecular weight Heparin, non-steroidal anti-inflammatory drugs, herbal supplements), for whom a dose interruption from Screening through 2-Months post-treatment (pre-treatment / treatment / biopsy phase) is contraindicated, are excluded from the study.
4. Any disorder (psychiatric, alcohol or substance abuse [within 12 months of treatment], physical disability) that might interfere with obtaining informed consent or the subject's ability to comply with study or protocol requirements, as determined by the Investigator.
5. Subjects who have used any tobacco product within 3 months prior to treatment.
6. Subjects previously treated with Apligraf®, Dermagraft or any other cell-based product, including autologous tissue at the treatment site.
7. Subjects who have received an investigational drug, device or biological/bioactive treatment within 30 days prior to treatment (medical or dental).
8. Subjects, who in the opinion of the Investigator, for any reason other than those listed above, will not be able to complete the study per protocol.
9. Subjects, as determined by Screening immunology testing, that have specific antibodies to VCT-01 donor cell human leukocyte antigens.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and changes from Baseline Immunology at 1, 3, 6 and 12 Months | Up to 12 months post-treatment
  Frequency and severity of reported adverse events and changes in results of immunology testing at Months 1, 3, 6 and 12 post-treatment as compared to baseline testing

SECONDARY OUTCOMES:
Healing parameter | Day 4 post-treatment
  Percentage area of questionable viability
Healing parameter | Day 14 post-treatment
  Percentage area of graft survival
Healing parameter | Up to 10 days post-treatment
  Histological and immunohistochemical analyses to examine cellular composition and tissue architecture.
Healing parameter | Up to 10 days post-treatment
  Microarray analysis to quantitatively measure molecular phenotypes expression.
Healing parameter | Up to 12 Months post-treatment
  Short tandem repeat analysis for persistence of VCT-01

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Tredget, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada